## Title: Bubble PEP Training Among Patient With Chronic Obstructive Pulmonary Disease in Pulmonary Function Effects

## **Statistical Analysis**

Principal Investigator: Szu-Yi Wang

ClinicalTrials.gov number: NCT04828837

2021/02/25

## **Statistical Analysis**

Statistical analyses were performed using the IBM statistical software SPSS Statistics version 22. The intention-to-treat analysis (ITT) method was employed for data analysis, and the expectation-maximization algorithm (EM) was used to handle missing data. We used t-tests for independent samples, and Fisher's exact tests when more than 20% of cells have expected frequencies <5 or less than 10 observations to examine the homogeneity between groups based on demographic characteristics. Descriptive statistics, including count, percentage, mean, and standard deviation, were used to summarize the data. The intervention effect was evaluated using the generalized estimating equation (GEE) statistical method. Two-tailed tests were conducted, and p-values less than .05 were considered statistically significant.